CLINICAL TRIAL: NCT05842954
Title: A Randomized, Open-label, Multicenter Study to Compare Efficacy, Safety and Tolerability of KLU156 With Coartem® in the Treatment of Uncomplicated Plasmodium Falciparum Malaria in Adults and Children Followed by an Extension Phase With Repeated KLU156 Treatment
Brief Title: Efficacy, Safety and Tolerability of KLU156 in Adults and Children With Uncomplicated P. Falciparum Malaria
Acronym: KALUMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Medicines for Malaria Venture (MMV), EDCTP, WANECAM (Unknown)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CKLU156A12301; 2022-002675-10 (EudraCT Number)
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Uncomplicated Plasmodium Falciparum Malaria
Keywords: malaria; Plasmodium falciparum; KLU156; Coartem; artemether; lumefantrine; ganaplacide
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The Novartis clinical trial team (CTT) will be blinded to the identity of the treatment from the time of randomization until the database lock for the analysis of the Core phase. Prior to unblinding the data of the Core phase (for the Novartis CTT), at least three DMC reviews are planned to minimize risks in this vulnerable patient population:
  1. Once the first 200 patients (across both treatment arms) in the Core phase have been dosed and followed up to at least Day 22.
  2. Once the first 750 patients (across both treatment arms) in the Core phase have been dosed and followed up to at least Day 22.
  3. Additional DMC reviews may be conducted ad-hoc during the study, as deemed necessary.
  All safety data from the Core phase as well as from the Extension phase that are available at these 2 scheduled timepoints will be included in the DMC reviews. After the database lock of the Core phase, the CTT will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KLU156 (Experimental): KLU156 once daily (QD) for 3 days under fed conditions (light meal).
  Interventions: Drug: KLU156
- Coartem (Active Comparator): Coartem twice a day (BID) for 3 days under fed conditions.
  Interventions: Drug: Coartem

INTERVENTIONS:
Drug: KLU156 — Oral use. KLU156 (400/480 mg) is the dose for patients with a bodyweight ≥ 35kg. Patients < 35kg will take a fraction of the dose according to weight group as defined in the protocol.
  Arms: KLU156
Drug: Coartem — Oral use. Dosing will be selected based on patient's body weight as per product's label.
  Arms: Coartem

SUMMARY:
This study aims to confirm the efficacy, safety and tolerability of KLU156, a fixed dose combination of ganaplacide (KAF156) and a solid dispersion formulation of lumefantrine (lumefantrine-SDF), when administered once daily for three days in adults and children ≥ 10 kg of body weight suffering from uncomplicated P. falciparum malaria (with or without other Plasmodium spp. co-infection).

In the Extension phase, the safety, tolerability and efficacy of repeated treatment with KLU156 will be assessed for a maximum of two years in patients who did not experience early treatment failure (ETF), who did not experience any study treatment-related SAE (Serious Adverse Event) previously and who gave informed consent to participate in the Extension phase.

DETAILED DESCRIPTION:
The purpose of this study is to confirm the efficacy, safety and tolerability of KLU156 in patients with uncomplicated P. falciparum malaria (with or without other Plasmodium spp. co-infection) by demonstrating that KLU156 is non-inferior to Coartem.

* The study duration will be 43 days (Core phase) plus up to 24 months (Extension phase).
* The treatment duration will be 3 days for each malaria episode.
* The visit frequency will be Days 1-3 (hospitalized) and 5 follow-up visits (Days 4, 8, 22, 29 and 43) in the Core phase and Days 1-3 (hospitalized) and 3 follow-up visits (Days 4, 8 and 29) in the Extension phase.

This study has two different primary outcomes depending on the submission (US New Drug Application (NDA) or non-US submissions).

ELIGIBILITY:
Key Inclusion criteria (Core phase)

1. Male or female patients ≥ 10 kg of body weight.
2. Microscopically confirmed diagnosis of uncomplicated P. falciparum malaria with an asexual P. falciparum parasitemia ≥ 1,000 and ≤ 200,000 parasites/µL at the time of pre-screening with or without other Plasmodium spp. co-infection.
3. Axillary temperature ≥ 37.5 ºC or oral temperature ≥ 38.0 ºC or tympanic/rectal temperature ≥ 38.5 ºC; or history of fever during the previous 24 hours (at least documented verbally)
4. Negative pregnancy test for patients of childbearing potential
5. Signed informed consent must be obtained before any assessment is performed; for minors, signed informed consent must be obtained from parent/legal guardian. If the parent/legal guardian is unable to read and write, then a witnessed consent according to local ethical standards is permitted. Patients who are capable of providing assent, must provide it along with parent/legal guardian consent or as per local ethical standards
6. The patient and/or their parent/legal guardian is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions and is likely to complete the study as planned.

Key Exclusion criteria (Core phase)

1. Signs and symptoms of severe malaria according to WHO 2015 (World Health Organization)
2. Concurrent febrile illnesses (e.g., typhoid fever, known or suspected dengue fever, known COVID19)
3. Severe malnutrition. For patients ≥ 12 years: body mass index (BMI) < 16.0. For children < 12 years: less than 70% of median normalized WHO reference weight or very low mid-upper arm circumference (MUAC < 115 mm)
4. Repeated vomiting (defined as > 3 times in the 24 hours prior to start of screening) or severe diarrhea (defined as > 3 watery stools in the 24 hours prior to start of screening)
5. Clinically relevant abnormalities of electrolyte balance which require correction, e.g., hypokalemia, hypocalcemia or hypomagnesemia
6. Anemia (hemoglobin level <7 g/dL)
7. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs (e.g., Human immunodeficiency virus (HIV) patients on antiretroviral therapy (ART) or tuberculosis (TB) patients on treatment), or which may jeopardize the patient in case of participation in the study.
8. Any of the following:

   * Aspartate Aminotransferase/ Alanine Aminotransferase (AST/ALT) > 3 x the upper limit of normal (ULN), regardless of the level of total bilirubin
   * Total bilirubin > 3 x ULN
   * Resting QT interval corrected by Fridericia's formula (QTcF) > 450 ms at screening
9. Prior antimalarial therapy or antibiotics with antimalarial activity within minimum of their five plasma half-lives (or within 4 weeks of screening if half-life is unknown)
10. History or family history of long QT syndrome or sudden cardiac death, or any other clinical condition known to prolong the QTc interval, such as history of symptomatic cardiac arrhythmias, clinically relevant bradycardia or severe heart disease
11. Pregnant or nursing (lactating) patients.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 2 Months to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1720 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
PCR-corrected adequate clinical and parasitological response (ACPR) | Day 29 (i.e., 28 days post-first dose administration)
  To confirm the efficacy of KLU156 in adults and children ≥ 10 kg of body weight suffering from uncomplicated malaria caused by P. falciparum (with or without other Plasmodium spp. co-infection) by demonstrating that KLU156 is non-inferior to Coartem (non-inferiority margin = 5%) based on the PCR-corrected ACPR at Day 29. This primary outcome is applicable to non-US submission.
Uncorrected ACPR (US NDA submission) | Day 29
  To further confirm the efficacy of KLU156 by demonstrating non-inferiority of KLU156 to Coartem (NI margin 7.5%) based on the uncorrected ACPR at Day 29. This primary outcome is applicable to US New Drug Application (NDA) submission.

SECONDARY OUTCOMES:
Uncorrected ACPR | Day 29
  To further confirm the efficacy of KLU156 by demonstrating non-inferiority of KLU156 to Coartem (NI margin 7.5%) based on the uncorrected ACPR at Day 29
PCR-corrected and uncorrected ACPR | Days 22 and 43 (i.e., 21 and 42 days post-first dose administration)
  To confirm the efficacy of KLU156 by assessing uncorrected and PCR-corrected ACPR at additional time points
Incidence rate of recrudescence and new infection | Days 22, 29 and 43
  Proportion of patients with recrudescence and new infections between the two treatment arms
Fever Clearance Time | Up to Day 3
  To confirm the efficacy of KLU156 by assessing fever clearance between the two treatment arms
Parasite Clearance Time | Up to Day 3
  To assess parasite clearance time between the two treatment arms
Gametocyte Clearance Time | Up to Day 3
  To confirm the efficacy of KLU156 by assessing gametocyte clearance between the two treatment arms
Proportion of patients with parasitemia | 12, 24, 48 and 72 hours after treatment
  For the parasitemia assessment, blood sampling can be done by means of a finger prick except when the timing for parasitology assessments coincides with time for clinical laboratory tests, in which case, blood sample can be taken from the venous blood collected for clinical laboratory analyses.
Gametocytemia | From baseline up to Day 43
  Disappearance or development of gametocytemia in patients with or without gametocytemia at baseline (pre-first dose administration), respectively
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 43
  Incidence and severity of AEs and SAEs by treatment group, including changes in vital signs, electrocardiograms (ECGs), and laboratory results qualifying and reported as AEs.
Extension phase: PCR-corrected and uncorrected ACPR | Day 29 of malaria episode
  To evaluate efficacy over repeated treatment with KLU156 in adults and children ≥ 10 kg of body weight suffering from uncomplicated malaria caused by P. falciparum (with or without other Plasmodium spp. co-infection) for a maximum of 2 years
Extension phase: KLU156-related AE/SAE incidence and severity by malaria episode | Up to 2 years
  To assess the safety and tolerability over repeated treatment with KLU156 in adults and children ≥ 10 kg of body weight suffering from uncomplicated malaria caused by P. falciparum (with or without other Plasmodium spp. co-infection) for a maximum of 2 years
Extension phase: Gametocyte carriage over time | Up to 2 years
  To assess gametocyte carriage over time by malaria episode in the extension phase

CONTACTS AND LOCATIONS:
Locations (32):
- Burkina Faso (5):
  - Novartis Investigative Site, Banfora
  - Novartis Investigative Site, Bobo-Dioulasso
  - Novartis Investigative Site, Nanoro
  - Novartis Investigative Site, Ouagadougou
  - Novartis Investigative Site, Sabou
- Côte d’Ivoire (3):
  - Novartis Investigative Site, Abidjan
  - Novartis Investigative Site, Agboville
  - Novartis Investigative Site, Azaguié
- Democratic Republic of the Congo (5):
  - Novartis Investigative Site, Kimpese, Bas-Congo Province
  - Novartis Investigative Site, Kisantu, Bas-Congo Province
  - Novartis Investigative Site, Lubumbashi, Du Haut Katanga
  - Novartis Investigative Site, Kenge, Kwango
  - Novartis Investigative Site, Masi-Manimba, Kwilu
- Gabon (2):
  - Novartis Investigative Site, Lambaréné
  - Novartis Investigative Site, Libreville
- Ghana (2):
  - Novartis Investigative Site, Kintampo
  - Novartis Investigative Site, Navrango
- Kenya (3):
  - Novartis Investigative Site, Kombewa
  - Novartis Investigative Site, Nairobi
  - Novartis Investigative Site, Siaya
- Novartis Investigative Site, Sotouba, Mali
- Novartis Investigative Site, Niamey, Niger
- Rwanda (4):
  - Novartis Investigative Site, Gicumbi, Northern Province
  - Novartis Investigative Site, Kigali
  - Novartis Investigative Site, Rubavu
  - Novartis Investigative Site, Rusizi
- Tanzania (3):
  - Novartis Investigative Site, Bagamoyo
  - Novartis Investigative Site, Korogwe Tanga
  - Novartis Investigative Site, Tanga
- Novartis Investigative Site, Tororo, Uganda
- Zambia (2):
  - Novartis Investigative Site, Nchelenge, Luapula Province
  - Novartis Investigative Site, Ndola

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.